CLINICAL TRIAL: NCT01711437
Title: EFFICACY, TOLERABILITY, AND SAFETY OF DIFFERENT BOWEL PREPARATIONS FOR COLONOSCOPY IN CHILDREN
Brief Title: Different Bowel Preparations for Colonoscopy In Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Giovanni Di Nardo, MD, Azienda Policlinico Umberto I
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: PEG-P2
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-10

CONDITIONS: Colonoscopy
Keywords: colonoscopy; colon cleansing; children; age 2 -18 years

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PEG-S (Experimental): polyethylene glycol 4000 solution with simethicon
  Interventions: Device: polyethylene glycol 4000 solution with simethicon
- PEG-CS + Bisacodyl (Experimental): PEG-CS is a new sulphate-free iso-osmotic formulation of PEG-4000 with citrates and simethicone
  Interventions: Device: PEG-4000 with citrates and simethicone
- PEG-ASC (Experimental): polyethylene glycol 3350 hyper-osmotic solution with ascorbic acid
  Interventions: Device: polyethylene glycol 3350 hyper-osmotic solution with ascorbic acid
- picoprep (Experimental): sodium picosulphate plus magnesium oxide and citric acid
  Interventions: Device: sodium picosulphate plus magnesium oxide and citric acid

INTERVENTIONS:
Device: PEG-4000 with citrates and simethicone — 1-4 bisacodyl 5-mg tablets (Lovoldyl) at 16:00, followed 2-3 hours later by 50 ml/kg (maximum 2 L) of PEG-CS solution. The patients were instructed to drink all solution in about 2-3 hours.
  Other Names: lovol-esse
  Arms: PEG-CS + Bisacodyl
Device: polyethylene glycol 4000 solution with simethicon — patients received a polyethylene glycol 4000 solution with simethicon (Selg Esse) starting at 3:00 p.m. the day before the colonoscopy at a dose of 100 ml/Kg (maximum 4 L). The patients were instructed to drink all solution in about 4-6 hours.
  Other Names: selg-esse
  Arms: PEG-S
Device: polyethylene glycol 3350 hyper-osmotic solution with ascorbic acid — patients received a polyethylene glycol 3350 hyper-osmotic solution with ascorbic acid (Moviprep) a dose of 50 ml/Kg (maximum 2 L) with 25 ml/kg additional clear fluid after completing solution intake.
  Other Names: moviprep
  Arms: PEG-ASC
Device: sodium picosulphate plus magnesium oxide and citric acid — patients received two sachets of sodium picosulphate plus magnesium oxide and citric acid (Picoprep), each diluted in 150 ml of water, at 14:00 and 6 hours later in the evening prior to the colonoscopy. Intake of at least 40-50 ml/kg of clear fluids
  Other Names: Picoprep
  Arms: picoprep

SUMMARY:
THE AIM OF THIS STUDY IS TO COMPARE THE EFFICACY, TOLERABILITY, AND SAFETY OF DIFFERENT BOWEL PREPARATIONS FOR COLONOSCOPY IN CHILDREN.

THE AIM OF THIS STUDY IS TO COMPARE THE OVERALL COLON CLEANSING

DETAILED DESCRIPTION:
COLONOSCOPY IS AN ESTABLISHED DIAGNOSTIC AND THERAPEUTIC TOOL IN A VARIETY OF GASTROINTESTINAL TRACT CONDITION AFFECTING CHILDREN AND ADOLESCENTs. FOR EXAMPLE: INFLAMMATORY BOWEL DISEASE, COLONIC POLYPS OR LOWER GASTROINTESTINAL TRACT BLEEDING.

THE IDEAL PREPARATION SHOULD BE OF LOW VOLUME, PALATABLE AND SUCCESSFUL IN COMPLETE COLON CLEANOUT.

PRIMARY AIMS OF THIS WERE TO COMPARE THE EFFICACY AND ACCEPTANCE OF FOUR METHODS OF BOWEL CLEANSING BEFORE COLONOSCOPY IN CHILDREN. SECONDARY AIMS WAS TO COMPARE THE SAFETY PROFILE OF THIS METHODS.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective colonoscopy in our Institution between 2 and 18 years of age were recruited for this study.

Exclusion Criteria:

1. requirement for urgent colonoscopy,
2. bowel obstruction,
3. known or suspected hypersensitivity to the active or other ingredients,
4. clinically significant electrolyte imbalance,
5. prior intestinal resection,
6. known metabolic, renal and cardiac disease

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy | During the performance of colonoscopy
  Preparation efficacy was evaluated by the blinded endoscopist according to the Boston Bowel Preparation scale (BBPS) consisting of four-point scoring system.
  The total score ranging from 0 to 9 was divided into four different classes: excellent cleansing (total score 8-9), good cleansing (total score 6-7), poor cleansing (total score 4-5) and inadequate cleansing (total score 0-3).

SECONDARY OUTCOMES:
safety | 4 days
  Adverse events were assessed on the day of colonoscopy by direct questioning and by telephone interview 48-96 hours after colonoscopy.
clinical tolerabiity | On the morning of colonoscopy, immediately before the procedure
  Tolerability assessment was based on the recording of occurrence and severity of GI symptoms such as nausea, bloating, abdominal, pain/cramps and anal discomfort
Compliance | On the morning of colonoscopy, immediately before the procedure
  Compliance was scored on a 3-point scale according to the percentage of drunk solution
Acceptability | On the morning of colonoscopy, immediately before the procedure
  The easiness of taking or swallowing the solution was graded according to the following scale: very severe distress = 4, severe distress = 3, moderate distress = 2, mild distress = 1, no distress = 0.

CONTACTS AND LOCATIONS:
Locations (1):
- Dipartimento di pediatria e neuropsichiatria Policlinico umberto l "università di roma la sapienza", Roma, Italy